CLINICAL TRIAL: NCT03937687
Title: The Effects of a Combination of TeaCrine®, Dynamine, and Caffeine on Marksmanship Accuracy and Reaction Time in ROTC Members, Military, and Law Enforcement Following a Mentally Fatiguing Protocol
Brief Title: The Effects of a Combination of TeaCrine®, Dynamine, and Caffeine in Law Enforcement
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of South Carolina (Other)
Collaborators: Compound Solutions Inc. (Industry); Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Shawn M. Arent, Principal Investigator, University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00096559
Record Dates: First submitted 2019-04-26; First posted 2019-05-06 (Actual); Last update posted 2021-09-30 (Actual); Status verified 2021-09

CONDITIONS: Caffeine, Teacrine, and Dynamine: Effects on Performance
MeSH Terms: interventions — Caffeine

STUDY DESIGN:
Intervention Model Description: Between-subjects, three condition groups
Who Masked: Participant, Investigator
Masking Description: Double-blind
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Placebo (Placebo Comparator): 300 mg cellulose
  Interventions: Drug: Placebo
- Caffeine (Experimental): 300 mg caffeine
  Interventions: Drug: Caffeine
- Caffeine Combination (Experimental): 150 mg caffeine with 100 mg Dynamine and 50 mg TeaCrine
  Interventions: Drug: Caffeine+TeaCrine+Dynamine

INTERVENTIONS:
Drug: Caffeine+TeaCrine+Dynamine — combination of caffeine, TeaCrine, and Dynamine
  Other Names: Combination
  Arms: Caffeine Combination
Drug: Placebo — Placebo
  Arms: Placebo
Drug: Caffeine — Caffeine
  Arms: Caffeine

SUMMARY:
The purpose of this randomized, placebo-controlled, three-condition, double-blind, between-subjects clinical trial is to determine and compare the effects of the combination of TeaCrine®, Dynamine, and caffeine to a placebo and caffeine condition on reaction time and target acquisition and accuracy. A secondary purpose is to observe the changes in hemodynamic variables in response to this combination.

DETAILED DESCRIPTION:
BASELINE ASSESSMENT:

* Subjects will report to the University of South Carolina Sport Science Lab normally hydrated and having refrained from eating for minimum 2 hours prior.
* Upon arrival, subjects will complete the informed consent and the Caffeine Frequency Questionnaire (CFQ) to assess their intake.
* Subjects will have body composition assessed using air displacement plethysmography (Bod Pod, Cosmed, Inc.) using standardized procedures.
* A salivary sample will be provided by each subject before beginning familiarization to analyze for presence of the CYP1A2 (caffeine) gene.
* Subjects will be familiarized with the cognitive testing protocols using the Dynavision D2TM board and TRAZER Sports Simulator. They will complete a shortened version of the mentally fatiguing condition on the DynavisionTM to familiarize with the protocol. They will be able to complete 3 trials of reaction time using the simulation on the TRAZER.
* Following this, subjects will then complete 3 trials of marksmanship assessment using the optical targetry system.

CONDITIONS:

* Following exercise familiarization, subjects will be randomly assigned to the condition of placebo (P), caffeine (C), or combination of caffeine + TeaCrine + Dynamine (DC). Sessions will be scheduled at the same time as the initial baseline/familiarization session.
* Subjects will be asked to maintain a normal sleep schedule in the week leading up to their session, maintaining the same wake time each day.
* Subjects will be asked to refrain from alcohol for 48 hours and caffeine 24 hours prior to their condition, with no major changes in food intake.
* Subjects will consume the supplement, complete the Multi-Component Training Distress Scale (MTDS) and will begin their session 30 minutes later.
* Sessions will include 30 minutes of a mentally fatiguing task on the Dynavision D2TM board, designed with a go/no-go stimulus. The blinds will be drawn and lights switched off to reduce glare on the board.
* At baseline and after each phase of the protocol, an assessment of psychological arousal will be taken using subjective measures of the Felt Arousal Scale (FAS) .
* Subjects will then perform the reaction time assessment on the TRAZER and shooting assessment. This will be performed twice. The TRAZER will consist of 40 targets, and the shooting assessment will be 8 shots with a tactical re-load followed by an additional 8 shots. A 2-minute rest will be taken between trials. Total time allotted for assessments will be 20 minutes.
* Subjects will then be seated in a room for 30 minutes, during which time they will read leisurely. At the completion of this time, subjects will complete the mentally fatiguing protocol once more (30 minutes). Following this, measures of reaction time and shooting assessment will be performed again (20 minutes).
* Heart rate will be monitored and recorded throughout testing to establish average and peak values during the reaction time and marksmanship tasks.
* Blood pressure will be measured pre- and post-testing using the Omron HEM 907XL Intellisense Pro Digital Blood Pressure cuff.

ELIGIBILITY:
Inclusion Criteria:

* Subject has provided written and dated informed consent to participate in the study.
* Subject is in good health as determined by physical examination and medical history.
* Subject is between the ages of 18 and 63.
* Subject is a current member of the military or law enforcement.

Exclusion Criteria:

* Subjects who have injuries that would prevent them from completing the protocol.
* Subjects who have migraine headaches.
* Subjects with a history of kidney or liver disease.
* Subjects with a history of caffeine sensitivity.
* Subjects currently taking OTC products containing pseudoephedrine or other stimulants.
* Subjects who drink more than four cups of coffee per day.

Ages: 18 Years to 63 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2019-05-04 (Actual); Primary Completion 2020-11-15 (Actual); Study Completion 2020-11-15 (Actual)

PRIMARY OUTCOMES:
Reaction time | 4 minutes, following the first 30-minute mental fatigue protocol
  Spatial reaction
Reaction time | 4 minutes, following the second 30-minute mental fatigue protocol
  Spatial reaction
Marksmanship | 2 minutes, following the first 30-minute mental fatigue protocol
  Simulated marksmanship using optical targetry
Marksmanship | 2 minutes, following the second 30-minute mental fatigue protocol
  Simulated marksmanship using optical targetry

SECONDARY OUTCOMES:
Blood pressure responses | 3 hours total
  Changes in blood pressure throughout the course of the protocol
Heart rate responses | 3 hours total
  Changes in heart rate throughout the course the protocol

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Rutgers University Center for Health and Human Performance, New Brunswick, New Jersey
  - University of South Carolina Sport Science Lab, Columbia, South Carolina

IPD SHARING:
Plan to Share IPD: No